CLINICAL TRIAL: NCT03831607
Title: A Phase 2, Open-label Phosphate Binder Switch Study of KHK7791 in Hyperphosphatemia Patients on Hemodialysis
Brief Title: A Phosphate Binder Switch Study of KHK7791 in Hyperphosphatemia Patients on HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7791-003
Record Dates: First submitted 2019-01-29; First posted 2019-02-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-04

CONDITIONS: Hyperphosphatemia
Keywords: Tenapanor; Hyperphosphatemia; Hemodialysis
MeSH Terms: conditions — Hyperphosphatemia | interventions — tenapanor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KHK7791 (Experimental): Patients start at KHK7791 30 mg BID and can down titrate weekly to 20, 15, 10, and 5 mg BID, sequentially based on a GI tolerability question.
  Interventions: Drug: KHK7791

INTERVENTIONS:
Drug: KHK7791 — KHK7791 30 mg, 20 mg ,10 mg or 5 mg tablets
  Other Names: Tenapanor

SUMMARY:
To evaluate the effect and safety of a switch from phosphate binders to KHK7791 to treat Hyperphosphatemia in patients on HD.

ELIGIBILITY:
Inclusion Criteria:

* Stable chronic renal failure patients who have undergone hemodialysis 3 times per week for at least 12 weeks until screening examination.
* Met certain conditions for dialysis excluding Dry Weight (Dialysate, Dialyzer, Frequency of Dialysis per Week, Dialysis Time, Blood Flow Rate, and Dialysate and Substitution Fluid Flow Rate) 2 weeks before screening examination.
* Taking at least 2 tablets of phosphate binder 3 times per day. The prescribed dosage regimen should have been unchanged for the period from 2 weeks before screening examination through pre-enrollment.
* Serum phosphorus levels should be between 3.5 and 7.0 mg/dL (inclusive) at screening examination.
* If on any vitamin D or calcimimetics regimen, the dosage regimen should have been unchanged for the last 2 weeks before screening examination.

Exclusion Criteria:

* iPTH > 600 pg/mL (should be based on the most recent value from patient's medical records before pre-enrollment)
* History of inflammatory bowel disease (IBD) or diarrhea predominant irritable bowel syndrome
* History of gastrectomy or enterectomy (excluding endoscopic resection and cecectomy) or having undergone gastrointestinal tract surgery within 3 months before screening examination.
* Severe heart disease (including congestive heart failure, defined as New York Heart Association [NYHA] cardiac functional classification of Class III or IV, and vascular lesions requiring hospitalization such as myocardial infarction), hepatic impairment (including AST/ALT ≥ 100 U/L before the start of observation period), or concurrent cirrhosis.
* Developed cerebrovascular disease (such as cerebral infarction and cerebral hemorrhage) or cardiovascular disease (such as acute myocardial infarction and unstable angina) requiring hospitalization within 6 months before screening examination.
* Uncontrollable hypertension or diabetes
* Scheduled for living donor kidney transplant, change in the mode of dialysis, home hemodialysis or plans to change the dialysis center (relocate to another hospital/clinic) during the study period.
* Any diagnosis of or treatment of malignancy within 5 years before screening examination (excluding basal cell carcinoma or surgically resected intraepithelial carcinoma of uterine cervix).

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who reduce the total number of taking phosphate binder tablets at the last assessment from baseline. | Week 26

SECONDARY OUTCOMES:
Serum phosphorus levels at each time point after the start of treatment | up to Week 26
Corrected serum calcium level at each time point after the start of treatment | up to Week 26

CONTACTS AND LOCATIONS:
Locations (1):
- Study Site 1, Niigata, Japan

IPD SHARING:
Plan to Share IPD: Undecided